CLINICAL TRIAL: NCT01835002
Title: Transcorneal Electrical Stimulation for the Treatment of Retinitis Pigmentosa - a Multicenter Safety Study of the Okustim ® System
Brief Title: Transcorneal Electrical Stimulation - Multicenter Safety Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Okuvision GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TESOLA
Record Dates: First submitted 2013-04-15; First posted 2013-04-18 (Estimated); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Retinitis Pigmentosa
Keywords: transcorneal electrostimulation
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OkuStim (Experimental): Electrostimulation Standard Treatment with OkuStim
  Interventions: Device: Transcorneal electrostimulation

INTERVENTIONS:
Device: Transcorneal electrostimulation — Weekly stimulation for 30 minutes with current of TES delivered of 150% of the individual phosphene threshold.
  Other Names: OkuStim; TES; TcES

SUMMARY:
The purpose of this study is to expand the safety assessment of repeated applications of an electrical current from a DTL-like electrode in patients with RP.

DETAILED DESCRIPTION:
This is a single-arm open label interventional safety trial with RP patients, who receive weekly TES for 6 months on 1 eye followed by observation for another 6 months without stimulation. The primary outcome measure is safety, indicated by the frequency and severity of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* patients with retinitis pigmentosa (rod-cone dystrophy) after prescription of electrical stimulation by an ophthalmologist
* adult patients who are capable of giving consent,
* Visual acuity ≥ 0.02
* because the electrode is to be positioned on the eye at home, the patient or his family members should have sufficient fine motor skills (assessment by the study physician)
* the patient must be capable of giving consent and a medical assessment that he/she is able to participate in the whole study according to the protocol

Exclusion Criteria:

* diabetic retinopathy
* neovascularisation of any origin
* after arterial or venous occlusion
* after retinal detachment
* silicone oil tamponade
* dry or exudative age-related macular degeneration
* macular edema
* all forms of glaucoma
* any form of corneal degeneration that reduces visual acuity
* systemic diseases that are difficult to control or manage, that could endanger the normal study schedule
* patients in a permanently poor general condition, which could hinder the regular attendance at control examinations in the clinic
* forms of mental illness related to the bipolar affective and schizoid-affective disorders, and all forms of dementia
* simultaneous participation in another interventional study or history of interventions whose effect may still persist

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2012-09; Primary Completion 2014-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
ophthalmic examinations | 6 months
  visual acuity slit lamp microscopy for examination of the anterior and posterior segment intraocular pressure measurement visual field examination Optical coherence tomography (OCT) Digital colour fundus photography

SECONDARY OUTCOMES:
Questionnaires | 6 months
  Questionnaires to collect the patient's perceived benefits of treatment and handling of the device

CONTACTS AND LOCATIONS:
Overall Officials: Florian Gekeler, Prof Dr med, Principal Investigator — Eberhard-Karls-Universität Tübingen
Locations (7):
- Glostrup Hospital and Kennedy Center, Glostrup Municipality, Denmark
- Germany (5):
  - University Eye Clinic Bonn, Bonn
  - Augenzentrum München, Munich
  - University Eye Clinic Regensburg, Regensburg
  - Zentrum für seltene Netzhauterkrankungen, AugenZentrum Siegburg, Siegburg
  - Centre for Ophthalmology at the eye clinic Tübingen, Tübingen
- Oslo University Hospital, Oslo, Norway

REFERENCES:
- [Background] Naycheva L, Schatz A, Rock T, Willmann G, Messias A, Bartz-Schmidt KU, Zrenner E, Gekeler F. Phosphene thresholds elicited by transcorneal electrical stimulation in healthy subjects and patients with retinal diseases. Invest Ophthalmol Vis Sci. 2012 Nov 1;53(12):7440-8. doi: 10.1167/iovs.12-9612. PMID 23049087
- [Background] Gekeler F; Arbeitsgruppe Elektrostimulation des Department fur Augenheilkunde am Universitats-Klinikum Tubingen. [Transcorneal electrostimulation]. Ophthalmologe. 2012 Feb;109(2):129-35. doi: 10.1007/s00347-011-2450-6. German. PMID 22350549
- [Background] Schatz A, Rock T, Naycheva L, Willmann G, Wilhelm B, Peters T, Bartz-Schmidt KU, Zrenner E, Messias A, Gekeler F. Transcorneal electrical stimulation for patients with retinitis pigmentosa: a prospective, randomized, sham-controlled exploratory study. Invest Ophthalmol Vis Sci. 2011 Jun 23;52(7):4485-96. doi: 10.1167/iovs.10-6932. PMID 21467183
- [Background] Schatz A, Arango-Gonzalez B, Fischer D, Enderle H, Bolz S, Rock T, Naycheva L, Grimm C, Messias A, Zrenner E, Bartz-Schmidt KU, Willmann G, Gekeler F. Transcorneal electrical stimulation shows neuroprotective effects in retinas of light-exposed rats. Invest Ophthalmol Vis Sci. 2012 Aug 15;53(9):5552-61. doi: 10.1167/iovs.12-10037. PMID 22807300
- [Background] Rock T, Schatz A, Naycheva L, Gosheva M, Pach J, Wilhelm B, Peters T, Bartz-Schmidt KU, Zrenner E, Willmann G, Gekeler F. [Effects of transcorneal electrical stimulation in patients with Stargardt's disease]. Ophthalmologe. 2013 Jan;110(1):68-73. doi: 10.1007/s00347-012-2749-y. German. PMID 23329121
- [Result] Jolly JK, Wagner SK, Martus P, MacLaren RE, Wilhelm B, Webster AR, Downes SM, Charbel Issa P, Kellner U, Jagle H, Ruther K, Bertelsen M, Bragadottir R, Prener Holtan J, van den Born LI, Sodi A, Virgili G, Gosheva M, Pach J, Zundorf I, Zrenner E, Gekeler F. Transcorneal Electrical Stimulation for the Treatment of Retinitis Pigmentosa: A Multicenter Safety Study of the OkuStim(R) System (TESOLA-Study). Ophthalmic Res. 2020;63(3):234-243. doi: 10.1159/000505001. Epub 2019 Nov 26. PMID 31775146